CLINICAL TRIAL: NCT00443586
Title: Age-27 Follow-up of Early Preventive Intervention
Brief Title: Follow-up Evaluation of Home Nurse Visitation Program for Socially Disadvantaged Women and Their Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-0002; R01MH070761 (NIH); DSIR 84-CTP
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Risk Reduction Behavior
Keywords: Nurse; Home Visitation; Welfare; Social Behavior
MeSH Terms: conditions — Risk Reduction Behavior; Social Behavior | interventions — Mass Screening; Transportation; Parturition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors were masked to original treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Developmental Screening (Active Comparator): Participants received sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age.
  Interventions: Behavioral: Developmental Screening
- Screening plus Transportation (Active Comparator): Participants received sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age; their mothers received free transportation for regular prenatal and well-child care (through child age two).
  Interventions: Behavioral: Developmental Screening; Behavioral: Screening plus Transportation
- Screening, Transport, Prenatal Visits (Active Comparator): Participants received sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age; their mothers received free transportation for regular prenatal and well-child care (through child age two), plus nurse home visiting during pregnancy.
  Interventions: Behavioral: Developmental Screening; Behavioral: Screening plus Transportation; Behavioral: Screening, Transport, Prenatal Visits
- Screen, Transport, Prenatal/Inf Visits (Experimental): Participants received regular sensory and developmental screening and referral for further evaluation and treatment of suspected problems at 12 and 24 months of age; their mothers received free transportation for regular prenatal and well-child care (through child age two), plus nurse home visiting during pregnancy and through child age two.
  Interventions: Behavioral: Developmental Screening; Behavioral: Screening plus Transportation; Behavioral: Screening, Transport, Prenatal Visits; Behavioral: Screen, Transport, Prenatal/Inf Visits

INTERVENTIONS:
Behavioral: Developmental Screening — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment at ages 12 and 24 months of age
Behavioral: Screening plus Transportation — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment at 12 and 24 months of age; their mothers were provided with free transportation for prenatal and well-child care through child age 2.
  Arms: Screen, Transport, Prenatal/Inf Visits; Screening plus Transportation; Screening, Transport, Prenatal Visits
Behavioral: Screening, Transport, Prenatal Visits — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment at 12 and 24 months of age; their mothers were provided with free transportation for prenatal and well-child care through child age 2, and were provided an average of 9 home visits by nurses during pregnancy.
  Arms: Screen, Transport, Prenatal/Inf Visits; Screening, Transport, Prenatal Visits
Behavioral: Screen, Transport, Prenatal/Inf Visits — Child participants were screened for sensory and developmental problems and referred for further evaluation and treatment at 12 and 24 months of age; their mothers were provided with free transportation for prenatal and well-child care through child age 2, and were provided an average of 9 home visits by nurses during pregnancy and 23 during the child's first two years of life.
  Arms: Screen, Transport, Prenatal/Inf Visits

SUMMARY:
This study will evaluate the long-term effects of a prenatal and early childhood home nurse visitation program for socially disadvantaged women and their children.

DETAILED DESCRIPTION:
Nearly half a million children are born each year to single, low-income mothers. Children born to socially disadvantaged mothers are more likely to experience chronic health problems, encounter child abuse and neglect, and receive insufficient health care. Home visitation by nurses during pregnancy and early childhood may prevent a wide range of health and developmental problems in children born to women who are either teenagers, unmarried, or of low economic status.

This study is associated with a home nurse visitation program that first began with 400 socially disadvantaged pregnant women between the years of 1977 and 1980 in an upstate New York semi-rural county. Participants in the original study were randomly assigned to participate in the home nurse visitation program or receive comparison services from pregnancy until the child's second birthday. Participants assigned to receive comparison services were provided with free transportation for prenatal and child care, as well as sensory and developmental screening for the child. Participants assigned to the home nurse visitation program were visited at home by a nurse 9 times during pregnancy and 23 times during the child's first 2 years of life. A follow-up study concluded that the home nurse visitation program reduced the number subsequent pregnancies, use of welfare, child abuse and neglect, and criminal behavior on the part of the socially disadvantaged mothers for up to 15 years after the birth of their first child.

This follow-up study will determine whether a home nurse visitation program has continued long-term effects on a child's health and development, 27 years later. Specifically, this study will evaluate whether the nurse-visited young adult offspring differ from the comparison group in their economic productivity; rates of child abuse and neglect; criminal behavior; mental health; abuse of substances; use of welfare, foster care, and healthcare in relation to government expenditures; and quality of their partnered relationships. Participants within the nurse-visited program group will be compared with each other to determine whether certain characteristics or factors, such as genetic vulnerabilities, environmental risks, or a history of child abuse, make someone less likely to benefit from a home nurse visitation program.

ELIGIBILITY:
Inclusion Criteria:

* Offspring of mothers who had participated in Elmira, N.Y. randomized clinical trial of prenatal and infant/toddler home visiting by nurses.
* Participants needed to be at least 27 years of age.

Ages: 27 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 345 (Estimated)
Dates: Start 2004-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Economic productivity (e.g., unemployment, employment in jobs with limited opportunities for career growth, use of welfare, rates of out-of-wedlock births) | Measured when child turns 27 years old
Quality of partnered relationships (violence, commitment, and communication) | Measured when child turns 27 years old
Rates of child abuse and neglect | Measured when child turns 27 years old
Rates of criminal behavior, arrests, convictions, and imprisonment | Measured when child turns 27 years old
Mental health and abuse of substances | Measured when child turns 27 years old
Government expenditures and higher tax revenues | Measured when child turns 27 years old

CONTACTS AND LOCATIONS:
Overall Officials: David L. Olds, PhD, Principal Investigator — University of Colorado, Denver; John Eckenrode, PhD, Study Director — Cornell University
Locations (1):
- Comprehensive Interdisciplinary Development Services (CIDS), Elmira, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data once the primary reports on this phase of the trial are published. This includes baseline data on maternal characteristics at registration during pregnancy and outcome data on primary outcomes for offspring participants at the 27-year follow-up. Data will be made available through the University of Michigan Inter-University Consortium for Political and Social Research (ICPSR). We anticipate archiving the data from this study with ICPSR by March 2018

REFERENCES:
- [Background] Izzo CV, Eckenrode JJ, Smith EG, Henderson CR, Cole R, Kitzman H, Olds DL. Reducing the impact of uncontrollable stressful life events through a program of nurse home visitation for new parents. Prev Sci. 2005 Dec;6(4):269-74. doi: 10.1007/s11121-005-0010-5. PMID 16075193
- [Background] Eckenrode J, Zielinski D, Smith E, Marcynyszyn LA, Henderson CR Jr, Kitzman H, Cole R, Powers J, Olds DL. Child maltreatment and the early onset of problem behaviors: can a program of nurse home visitation break the link? Dev Psychopathol. 2001 Fall;13(4):873-90. PMID 11771912
- [Background] Eckenrode J, Ganzel B, Henderson CR Jr, Smith E, Olds DL, Powers J, Cole R, Kitzman H, Sidora K. Preventing child abuse and neglect with a program of nurse home visitation: the limiting effects of domestic violence. JAMA. 2000 Sep 20;284(11):1385-91. doi: 10.1001/jama.284.11.1385. PMID 10989400
- [Background] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R. Intellectual impairment in children of women who smoke cigarettes during pregnancy. Pediatrics. 1994 Feb;93(2):221-7. PMID 8121734
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R. Prevention of intellectual impairment in children of women who smoke cigarettes during pregnancy. Pediatrics. 1994 Feb;93(2):228-33. PMID 7510063
- [Background] Olds DL, Henderson CR Jr, Kitzman H. Does prenatal and infancy nurse home visitation have enduring effects on qualities of parental caregiving and child health at 25 to 50 months of life? Pediatrics. 1994 Jan;93(1):89-98. PMID 8265329
- [Background] Olds DL, Henderson CR Jr, Phelps C, Kitzman H, Hanks C. Effect of prenatal and infancy nurse home visitation on government spending. Med Care. 1993 Feb;31(2):155-74. doi: 10.1097/00005650-199302000-00006. PMID 8433578
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R, Chamberlin R. Improving the life-course development of socially disadvantaged mothers: a randomized trial of nurse home visitation. Am J Public Health. 1988 Nov;78(11):1436-45. doi: 10.2105/ajph.78.11.1436. PMID 3052116
- [Background] Olds DL, Henderson CR Jr, Chamberlin R, Tatelbaum R. Preventing child abuse and neglect: a randomized trial of nurse home visitation. Pediatrics. 1986 Jul;78(1):65-78. PMID 2425334